CLINICAL TRIAL: NCT06031896
Title: The Comparison of the Severity of Periodontitis at the Buccal and Palatal Site
Brief Title: The Severity of Periodontitis at the Buccal and Palatal Site
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: The Dental Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-116
Record Dates: First submitted 2023-09-04; First posted 2023-09-11 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Periodontal Diseases
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No interventions — No interventions

SUMMARY:
To record and compare the periodontal conditions of buccal and palatal sites in patients

ELIGIBILITY:
Inclusion Criteria:

* patients with diagnosed periodontitis

Exclusion Criteria:

* compromised systematic health (uncontrolled hypertension, diabetes, impaired bone metabolism condition, etc.), uncontrolled periodontal disease, smoking > 20 cigarettes/day or recent chemotherapy/radiotherapy in the oral and maxillofacial regions

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: As many patients as investigators can collect
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
probing depth | 3 years
  the probing depth of buccal and palatal sites of teeth in one patient

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of Stomatology, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China